CLINICAL TRIAL: NCT00965419
Title: Long-Term, Open-Label, Safety Study of LY2216684 in Pediatric Patients With Attention Deficit/Hyperactivity Disorder
Brief Title: A Study of Pediatric Participants With Attention Deficit/Hyperactivity Disorder
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Terminated due to low 5 year completer number and not meeting primary objective.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11332; H9P-MC-LNDH (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Results first posted 2018-04-27 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Edivoxetine (Experimental): All enrolled participants were administered starting dose of 0.1 milligram per kilogram per day (mg/kg/day), or participant specific known stable dose, rollover participants (LNBJ [No NCT number]) and (LNBF [NCT00922636]), up to 0.3 mg/kg/day, oral, daily for up to 5 years.
  Interventions: Drug: Edivoxetine

INTERVENTIONS:
Drug: Edivoxetine — 0.1 mg/kg/day or participant specific known stable dose, rollover participants (LNBJ [No NCT number]) and (LNBF [NCT00922636]), up to 0.3 mg/kg/day, oral, daily for up to 5 years.
  Other Names: LY2216684

SUMMARY:
The primary purpose of the study is to assess long-term safety and tolerability of Edivoxetine in pediatric participants with attention deficit hyperactive disorder (ADHD).

ELIGIBILITY:
INCLUSION CRITERIA:

-Participants must meet Diagnostic and Statistical Manual of Mental Disorders 4th Ed (DSM-IV) diagnostic criteria for ADHD (inattentive, hyperactive/impulsive, or combined subtypes) based on an interview by an experienced clinician and confirmed using the Kiddie Schedule for Affective Disorders and Schizophrenia for School Aged Children-Present (SADS) and Lifetime Version (K-SADS-PL) at Visit 1 for new participants and in the parent trial for rollover participants.

-Participants must have an ADHDRS-IV-Parent: Inv total score of at least 1.5 standard deviations above the age/gender norm at both screening/randomization. New participants must have a Clinical Global Impressions-Attention-Deficit/Hyperactivity Disorder- Severity (CGI-ADHD-S) score greater than or equal to 4 at both screening/randomization.

* Participants of child-bearing potential agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug. Female participants of child-bearing potential must test negative for pregnancy at the time of enrollment based on a urine pregnancy test.
* Participants must have laboratory results, showing no clinically significant abnormalities.
* Parents/participants must have a degree of understanding sufficient to communicate suitably with the investigator/ study coordinator.
* Participants must be of normal intelligence.
* Participants/parents must have been judged by the investigator to be reliable to keep appointments for clinic visits/all tests, including venipunctures and examinations required by the protocol.
* Participants must be able to swallow tablets.

EXCLUSION CRITERIA:

* Participants who weigh less than 16 kg at screening/randomization.
* Female participants who are pregnant/breastfeeding.
* Participants who have previously withdrawn/discontinued early from this study or any other study investigating Edivoxetine.
* Participants who have a history of Bipolar I/II disorder, psychosis, or pervasive developmental disorder.
* Participants with a history of any seizure disorder or known electroencephalographic (EEG) abnormalities in the absence of seizures.
* Participants who are at serious suicidal risk.
* Participants with a history of severe allergies to more than 1 class of medications, or multiple adverse drug reactions, or known hypersensitivity to Edivoxetine.
* Participants with a history of alcohol or drug abuse/dependence within the past 3 months of screening, or who are currently using alcohol, drugs of abuse, or any prescribed or over-the-counter medication in a manner that the investigator considers indicative of abuse/dependence.
* Participants who screen positive for drugs of abuse cannot participate.
* Participants who have a medical condition that would increase sympathetic nervous system activity markedly, or who are taking a medication on a daily basis that has sympathomimetic activity are excluded.
* Participants with problems that would be exacerbated by increased norepinephrine tone including a history of cardiovascular disease, thyroid dysfunction, glaucoma, or urinary retention.
* Participants who at any time during the study are likely to need psychotropic medications apart from the drugs under study.
* Participants who have used a monoamine oxidase inhibitor (MAOI) during the 2 weeks prior to randomization.
* Participants with current or past history of clinically significant hypertension.
* Participants who are currently enrolled in, or discontinued within the last 30 days from a clinical trial involving an off-label use of an investigational drug, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Participants whose family anticipates a move outside the geographic range of the investigative site during participation in the study or who plan extended travel inconsistent with the recommended visit intervals.
* Participants who, in the opinion of the investigator, are unsuitable in any other way to participate in this study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 267 (Actual)
Dates: Start 2009-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (19):
- United States (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spring Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., University Park, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Smyrna, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Libertyville, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester Hills, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Jackson, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lubbock, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herndon, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kelowna, British Columbia, Canada
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santurce, Puerto Rico
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuei Shan Hsiang, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants that received edivoxetine during the open-label treatment phase for up to 5 years and follow-up phase.
Groups:
- Edivoxetine: Edivoxetine: 0.1 milligram (mg)/kilogram (kg)/day or participant specific known stable dose, rollover participants (LNBJ [No NCT number]) and (LNBF [NCT00922636]), up to 0.3 mg/kg/day, oral, daily for up to 5 years.
Period: Open Label Treatment for Responders
Arm/Group | Edivoxetine
Started | 267
Not Lost to f/u at First Post-baseline | 264
Completed | 20
Not Completed | 247
Not completed — Adverse Event | 33
Not completed — Entry Criteria Not Met | 1
Not completed — Protocol Violation | 21
Not completed — Withdrawal by Subject | 27
Not completed — Physician Decision | 6
Not completed — Sponsor Decision | 5
Not completed — Parent/Caregiver Decision | 41
Not completed — Lack of Efficacy | 67
Not completed — Lost to Follow-up | 46
Period: Follow-up Phase
Arm/Group | Edivoxetine
Started (Participants who dropped out of treatment period early had the option to enter follow-up period.) | 80
Completed | 18
Not Completed | 62
Not completed — Adverse Event | 9
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 8
Not completed — Physician Decision | 4
Not completed — Parent/Caregiver Decision | 9
Not completed — Lack of Efficacy | 28

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Edivoxetine: 0.1 mg/kg/day or participant specific known stable dose (rollover participants) up to 0.3 mg/kg/day, oral, daily for up to 5 years.
Arm/Group | All Participants
Number analyzed (Participants) | 267
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.64 (2.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 65
  Not Hispanic or Latino | 202
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 60
  White | 180
  More than one race | 14
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 9
  Puerto Rico | 11
  United States | 235
  Taiwan | 10
  Mexico | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With At Least One Serious Adverse Events (SAE) Over the Duration of the Study
Description: Percentage of Participants experienced at least one SAE during the study. A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline Through Week 252
Population: All enrolled participants who did not discontinue from the study for the reason 'Lost to follow up' at the first post-baseline observation and who had baseline and at least one post-baseline SAE assessment.
Measure: Number; unit: percentage of participants
Groups:
- Edivoxetine: Edivoxetine: 0.1 mg/kg/day or participant specific known stable dose (rollover participants) up to 0.3 mg/kg/day, oral, daily for up to 5 years.
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
percentage of participants | 2.65

2. Primary Outcome: Number of Participants With At Least One SAE
Description: Number of Participants experienced at least one SAE during the study. A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline Through Week 252
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
Participants | 7

3. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Percentage of Participants had at least one TEAE during the study. A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline Through Week 252
Population: All enrolled participants who did not discontinue from the study for the reason 'Lost to follow up' at the first post-baseline observation and who had baseline and at least one post-baseline TEAE assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
percentage of participants | 76.89

4. Secondary Outcome: Number of Participants With At Least One TEAE
Description: Number of participants had at least one TEAE during the study. A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline Through Week 252
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
Participants | 203

5. Secondary Outcome: Percentage of Participants With Discontinuation Due to Adverse Events (DCAEs)
Time Frame: Baseline Through Week 252
Population: All enrolled participants who did not discontinue from the study for the reason 'Lost to follow up' at the first post-baseline observation.
Measure: Number; unit: percentage of participants
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
percentage of participants | 12.50

6. Secondary Outcome: Number of Participants With At Least One DCAEs
Time Frame: Baseline Through Week 252
Population: All enrolled participants who did not discontinue from the study for the reason 'Lost to follow up' at the first post-baseline observation and who had baseline and at least one post-baseline DCAE assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
Participants | 33

7. Secondary Outcome: Percentage of Participants Who Discontinued Due to Any Reason
Time Frame: Baseline Through Week 252
Population: All enrolled participants who had evaluable discontinuation data.
Measure: Number; unit: Percentage of participants
Arm/Group | Edivoxetine
Number analyzed (Participants) | 267
Percentage of participants | 92.51

8. Secondary Outcome: Number of Participants Who Discontinued Due to Any Reason
Time Frame: Baseline Through Week 252
Population: All enrolled participants who had evaluable discontinuation data.
Measure: Count of Participants; unit: Participants
Arm/Group | Edivoxetine
Number analyzed (Participants) | 267
Participants | 247

9. Secondary Outcome: Percentage of Participants With Columbia-Suicide Severity Rating Scale (CSSRS) for Each Category
Description: Percentage of Participants in each category of CSSRS captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. Participants with suicidal ideation were those who had yes to any of the following questions: Wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intent to act, active suicidal ideation with some intent to act, without specific plan, and active suicidal ideation with specific plan and intent. Suicidal behavior included those who had yes to any of the following questions: Preparatory acts or behavior, Aborted attempt, Interrupted attempt, Non-fatal suicide attempt, Completed suicide.
Time Frame: Baseline Through Week 252, Baseline, 1-month (mo) Follow-Up (f/u)
Population: All enrolled participants who did not discontinue from the study for the reason 'Lost to follow up' at the first post-baseline observation and who had baseline and at least one post-baseline CSSRS assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
percentage of participants
  0-5 Years (Suicidal Ideation) | 5.68
  0-5 Years (Suicidal Behavior) | 0.00
  0-5 Yrs (Non-suicidal self-injurious) | 0.38
  1 month f/u (Suicidal Ideation): number analyzed (Participants) | 79
  1 month f/u (Suicidal Ideation) | 1.27
  1 month f/u (Suicidal Behavior): number analyzed (Participants) | 79
  1 month f/u (Suicidal Behavior) | 0.00
  1 mo f/u (Non-suicidal self-injurious behavior): number analyzed (Participants) | 79
  1 mo f/u (Non-suicidal self-injurious behavior) | 0.00

10. Secondary Outcome: Mean Change From Baseline Z-scores for Height
Description: A z-score is the number of standard deviations a data point is from the mean. Z-scores range from -3 standard deviations (far left of the mean in normal distribution curve) up to +3 standard deviations (far right of the mean in normal distribution curve).
Time Frame: Baseline, Week 60; Baseline, Week 240
Population: All enrolled participants who did not discontinue from the study for the reason 'Lost to follow up' at the first post-baseline observation and who had baseline and at least one post-baseline Z-score assessment.
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
Z-Score
  Week 60: number analyzed (Participants) | 104
  Week 60 | -0.05 (0.36)
  Week 240: number analyzed (Participants) | 24
  Week 240 | -0.11 (0.53)

11. Secondary Outcome: Mean Change From Baseline Z-Score for Weight
Description: as for outcome 10
Time Frame: Baseline, Week 60; Baseline, Week 240
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
Z-Score
  Week 60: number analyzed (Participants) | 104
  Week 60 | -0.17 (0.37)
  Week 240: number analyzed (Participants) | 24
  Week 240 | -0.25 (0.77)

12. Secondary Outcome: Mean Change From Baseline Z-Score in Body Mass Index (BMI)
Time Frame: Baseline, Week 60; Baseline, Week 240
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
Z-Score
  Week 60: number analyzed (Participants) | 104
  Week 60 | -0.20 (0.40)
  Week 240: number analyzed (Participants) | 24
  Week 240 | -0.32 (0.83)

13. Secondary Outcome: Percentage of Participants With Response Rates
Time Frame: Week 12
Population: Zero participants were analyzed for this outcome measure, due to all participants being roll-over from two previous edivoxetine trials (LNBJ [No NCT number]) and (LNBF [NCT00922636])This outcome measure and analysis was not applicable to roll-over participants.
Arm/Group | Edivoxetine
Number analyzed (Participants) | 0

14. Secondary Outcome: Number of Participants With a Response Rate
Time Frame: Week 12
Population: Zero participants were analyzed for this outcome measure. Data was not collected for this outcome for participants due to all participants being roll-over from two previous edivoxetine trials (LNBJ [No NCT number]) and (LNBF [NCT00922636]). This outcome measure was not applicable to roll-over participants.
Arm/Group | Edivoxetine
Number analyzed (Participants) | 0

15. Secondary Outcome: Survival Curve Time to Response
Time Frame: Week 12
Population: as for outcome 14
Arm/Group | Edivoxetine
Number analyzed (Participants) | 0

16. Secondary Outcome: Percentage of Participants in Sexual Maturation on Tanners Scale
Description: Participant's stage of sexual maturation were assessed using the Tanner staging measure for determining pubertal development in male and female participants. Tanner staging includes a self-assessment of pubic hair development (both males and females), genital development (males), and breast development (females). Tanner stage (pubic) is a score of range 1-5 where 1=no development and 5=adult pubic hair. Tanner stage (breast) is a score of range 1-5 where 1=no development and 5=adult breast. Tanner stages (1-5) were used to characterize physical development in children, adolescents, and adults. The stages were based on external primary and secondary sex characteristics, such as the size of the breasts, genitalia, and development of pubic hair. Tanner stage is considered going up when the organs grow bigger.
Time Frame: Baseline Up to Week 252
Population: All enrolled participants who did not discontinue from the study for the reason 'Lost to follow up' at the first post-baseline observation and who had baseline and at least one post-baseline Tanners scale assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
percentage of participants
  Pubic Hair Male Tanner I: number analyzed (Participants) | 100
  Pubic Hair Male Tanner I | 25.00
  Pubic Hair Male Tanner II: number analyzed (Participants) | 100
  Pubic Hair Male Tanner II | 11.00
  Pubic Hair Male Tanner III: number analyzed (Participants) | 100
  Pubic Hair Male Tanner III | 10.00
  Pubic Hair Male Tanner IV: number analyzed (Participants) | 100
  Pubic Hair Male Tanner IV | 23.00
  Pubic Hair Male Tanner V: number analyzed (Participants) | 100
  Pubic Hair Male Tanner V | 31.00
  Pubic Hair Female Tanner I: number analyzed (Participants) | 48
  Pubic Hair Female Tanner I | 12.50
  Pubic Hair Female Tanner II: number analyzed (Participants) | 48
  Pubic Hair Female Tanner II | 14.58
  Pubic Hair Female Tanner III: number analyzed (Participants) | 48
  Pubic Hair Female Tanner III | 6.25
  Pubic Hair Female Tanner IV: number analyzed (Participants) | 48
  Pubic Hair Female Tanner IV | 20.83
  Pubic Hair Female Tanner V: number analyzed (Participants) | 48
  Pubic Hair Female Tanner V | 45.83
  Genital Development Male Tanner I: number analyzed (Participants) | 100
  Genital Development Male Tanner I | 22.00
  Genital Development Male Tanner II: number analyzed (Participants) | 100
  Genital Development Male Tanner II | 11.00
  Genital Development Male Tanner III: number analyzed (Participants) | 100
  Genital Development Male Tanner III | 18.00
  Genital Development Male Tanner IV: number analyzed (Participants) | 100
  Genital Development Male Tanner IV | 17.00
  Genital Development Male Tanner V: number analyzed (Participants) | 100
  Genital Development Male Tanner V | 32.00
  Breast Development Female Tanner I: number analyzed (Participants) | 48
  Breast Development Female Tanner I | 16.67
  Breast Development Female Tanner II: number analyzed (Participants) | 48
  Breast Development Female Tanner II | 6.25
  Breast Development Female Tanner III: number analyzed (Participants) | 48
  Breast Development Female Tanner III | 16.67
  Breast Development Female Tanner IV: number analyzed (Participants) | 48
  Breast Development Female Tanner IV | 22.92
  Breast Development Female Tanner V: number analyzed (Participants) | 48
  Breast Development Female Tanner V | 37.50

17. Secondary Outcome: Number of Participants in Sexual Maturation on Tanners Scale
Description: as for outcome 16
Time Frame: Baseline Up to Week 252
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
Participants
  Pubic Hair Male Tanner I: number analyzed (Participants) | 100
  Pubic Hair Male Tanner I | 25
  Pubic Hair Male Tanner II: number analyzed (Participants) | 100
  Pubic Hair Male Tanner II | 11
  Pubic Hair Male Tanner III: number analyzed (Participants) | 100
  Pubic Hair Male Tanner III | 10
  Pubic Hair Male Tanner IV: number analyzed (Participants) | 100
  Pubic Hair Male Tanner IV | 23
  Pubic Hair Male Tanner V: number analyzed (Participants) | 100
  Pubic Hair Male Tanner V | 31
  Pubic Hair Female Tanner I: number analyzed (Participants) | 48
  Pubic Hair Female Tanner I | 6
  Pubic Hair Female Tanner II: number analyzed (Participants) | 48
  Pubic Hair Female Tanner II | 7
  Pubic Hair Female Tanner III: number analyzed (Participants) | 48
  Pubic Hair Female Tanner III | 3
  Pubic Hair Female Tanner IV: number analyzed (Participants) | 48
  Pubic Hair Female Tanner IV | 10
  Pubic Hair Female Tanner V: number analyzed (Participants) | 48
  Pubic Hair Female Tanner V | 22
  Genital Development Male Tanner I: number analyzed (Participants) | 100
  Genital Development Male Tanner I | 22
  Genital Development Male Tanner II: number analyzed (Participants) | 100
  Genital Development Male Tanner II | 11
  Genital Development Male Tanner III: number analyzed (Participants) | 100
  Genital Development Male Tanner III | 18
  Genital Development Male Tanner IV: number analyzed (Participants) | 100
  Genital Development Male Tanner IV | 17
  Genital Development Male Tanner V: number analyzed (Participants) | 100
  Genital Development Male Tanner V | 32
  Breast Development Female Tanner I: number analyzed (Participants) | 48
  Breast Development Female Tanner I | 8
  Breast Development Female Tanner II: number analyzed (Participants) | 48
  Breast Development Female Tanner II | 3
  Breast Development Female Tanner III: number analyzed (Participants) | 48
  Breast Development Female Tanner III | 8
  Breast Development Female Tanner IV: number analyzed (Participants) | 48
  Breast Development Female Tanner IV | 11
  Breast Development Female Tanner V: number analyzed (Participants) | 48
  Breast Development Female Tanner V | 18

18. Secondary Outcome: Percentage of Participants With Tobacco, Alcohol and Marijuana Use
Time Frame: Week 60 through Week 252
Population: All enrolled participants who did not discontinue from the study for the reason 'Lost to follow up' at the first post-baseline observation and who had baseline and at least one post-baseline tobacco, alcohol, and marijuana use assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
percentage of participants
  Current Tobacco Use Week 60: number analyzed (Participants) | 104
  Current Tobacco Use Week 60 | 0
  Current Alcohol Use Week 60: number analyzed (Participants) | 104
  Current Alcohol Use Week 60 | 0
  Current Marijuana Use Week 60: number analyzed (Participants) | 104
  Current Marijuana Use Week 60 | 0
  Current Tobacco Use Week 252: number analyzed (Participants) | 20
  Current Tobacco Use Week 252 | 0
  Current Alcohol Use Week 252: number analyzed (Participants) | 20
  Current Alcohol Use Week 252 | 0
  Current Marijuana Use Week 252: number analyzed (Participants) | 20
  Current Marijuana Use Week 252 | 0

19. Secondary Outcome: Number of Participants With Tobacco, Alcohol and Marijuana Use
Time Frame: Week 60 through Week 252
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
Participants
  Current Tobacco Use Week 60: number analyzed (Participants) | 104
  Current Tobacco Use Week 60 | 0
  Current Alcohol Use Week 60: number analyzed (Participants) | 104
  Current Alcohol Use Week 60 | 0
  Current Marijuana Use Week 60: number analyzed (Participants) | 104
  Current Marijuana Use Week 60 | 0
  Current Tobacco Use Week 252: number analyzed (Participants) | 20
  Current Tobacco Use Week 252 | 0
  Current Alcohol Use 252: number analyzed (Participants) | 20
  Current Alcohol Use 252 | 0
  Current Marijuana Use Week 252: number analyzed (Participants) | 20
  Current Marijuana Use Week 252 | 0

20. Secondary Outcome: Mean Change From Baseline of Each Score Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version: Investigator Administered and Scored (ADHDRS-IV-Parent:Inv) (Hyperactive/Impulsive, Inattentive and Total Score)
Description: The ADHDRS-IV-Parent scale measures the 18 symptoms contained in the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) diagnosis of Attention-Deficit/Hyperactivity Disorder. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total score is computed as the sum of the 18 items and ranges from 0 to 54. Inattention and Hyperactivity-Impulsivity subscales consisted of 9 items each, for total subscale scores ranging from 0 to 27. Higher total and subscale scores are indicative of more severe symptoms. Least-squares (LS) mean change from baseline was adjusted for repeated measure analysis included baseline score and visit time in the model.
Time Frame: Baseline, Week 12; Baseline, Week 60; Baseline, Week 252
Population: All enrolled participants who did not discontinue from the study for the reason 'Lost to follow up' at the first post-baseline observation and who had baseline and at least one post-baseline ADHDRS-IV-Parent assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
units on a scale
  Hyperactivity Impulsivity subscale Week 12: number analyzed (Participants) | 207
  Hyperactivity Impulsivity subscale Week 12 | -3.45 (0.33)
  Hyperactivity Impulsivity subscale Week 60: number analyzed (Participants) | 102
  Hyperactivity Impulsivity subscale Week 60 | -4.27 (0.38)
  Hyperactivity Impulsivity subscale Week 252: number analyzed (Participants) | 20
  Hyperactivity Impulsivity subscale Week 252 | -7.48 (0.46)
  Inattention Score Week 12: number analyzed (Participants) | 207
  Inattention Score Week 12 | -3.91 (0.38)
  Inattention Score Week 60: number analyzed (Participants) | 102
  Inattention Score Week 60 | -3.69 (0.45)
  Inattention Score Week 252: number analyzed (Participants) | 20
  Inattention Score Week 252 | -5.59 (0.73)
  Total Score Week 12: number analyzed (Participants) | 207
  Total Score Week 12 | -7.28 (0.65)
  Total Score Week 60: number analyzed (Participants) | 102
  Total Score Week 60 | -7.83 (0.76)
  Total Score Week 252: number analyzed (Participants) | 20
  Total Score Week 252 | -12.82 (1.06)

21. Secondary Outcome: Mean Change From Baseline of Total Score Clinical Global Impressions-Attention-Deficit/Hyperactivity Disorder-Severity (CGI-ADHD-S)
Description: The CGI-ADHD-S measures severity of the participants overall severity of ADHD symptoms. The score ranges from 1 to 7 (1=normal, not at all ill; 7=among the most extremely ill participants). LS mean change from baseline was adjusted for repeated measure analysis included baseline score and visit time in the model.
Time Frame: Baseline, Week 12; Baseline, Week 60; Baseline, Week 252
Population: All enrolled participants who did not discontinue from the study for the reason 'Lost to follow up' at the first post-baseline observation and who had baseline and at least one post-baseline CGI-ADHD-S assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
units on a scale
  Week 12: number analyzed (Participants) | 207
  Week 12 | -0.73 (0.07)
  Week 60: number analyzed (Participants) | 103
  Week 60 | -0.85 (0.10)
  Week 252: number analyzed (Participants) | 20
  Week 252 | -0.97 (0.17)

22. Secondary Outcome: Mean Change of Total Score Teacher-rated Swanson Nolan, and Pelham Rating Scale-Revised (SNAP-IV) ADHD Subscales (Hyperactive/Impulsive, Inattentive and Total Score)
Description: The SNAP-IV is a revision of the Swanson, Nolan, and Pelham (SNAP) Questionnaire (Swanson et al 1983). The SNAP-IV: ADHD Inattention Subscale (items 1-9) scores the intensity of each item during the last seven days on a 0 to 3 scale (0=not at all, 1=just a little, 2=pretty much, 3=very much). Possible scores range from 0-27. Lower scores indicate a lesser intensity of inattention and higher scores a greater intensity. The SNAP-IV ADHD Hyperactivity/Impulsivity Subscale (items 10-18) scores the intensity of each item in the last seven days on a 0 to 3 scale (0=not at all, 1=just a little, 2=pretty much, 3=very much). Possible scores range from 0-27. Lower scores indicate a lesser intensity of hyperactivity/impulsivity and higher scores, a greater intensity. SNAP-IV ADHD Combined Scale score (inattention + hyperactivity/impulsivity) ranges from 0-54. A low score of 0 indicates less inattention + hyperactivity/impulsivity. A high score of 54 indicates more inattention + hyperactivity.
Time Frame: Baseline, Week 12
Population: All enrolled participants with baseline and at least one post-baseline SNAP-IV assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edivoxetine
Number analyzed (Participants) | 14
units on a scale
  Inattention Score | 0.04 (0.42)
  Hyperactivity/Impulsivity Score | 0.05 (0.38)
  Total Score | 0.04 (0.32)

23. Secondary Outcome: Mean Change From Baseline of Total Score SNAP-IV Oppositional Defiant Disorder (ODD) Subscale
Description: The SNAP-IV ODD subscale includes items #21 to #28. Each item is scored on a 0 to 3 scale (0 = "Not At All", 1 = "Just A Little", 2 = "Pretty Much", 3 = "Very Much"). Score ranges from 0-24. The lowest possible score is 0; highest is 24. Higher scores indicate a greater presence of ODD and lowers scores a lower presence of ODD.
Time Frame: Baseline, Week 12
Population: All enrolled participants with baseline and at least one post-baseline SNAP-IV assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edivoxetine
Number analyzed (Participants) | 14
units on a scale | 0.02 (0.23)

24. Secondary Outcome: Mean Change From Baseline of Each Total Score Conners Comprehensive Behavior Rating Scales (CP-CBRS) Diagnostic and Statistical Manual of Mental Disorders, 4th Ed, Text Revision (DSM-IV-TR) for Symptom Subscales Manic Episode and Mixed Episode
Description: The Conners CBRS measures behaviors, emotions, and academic problems in children and adolescents. DSM-IV-TR symptom scales is included and assesses the following disorders: ADHD, conduct disorder, ODD, major depressive episode, manic episode, mixed episode, generalized anxiety disorder, separation anxiety disorder, social phobia, obsessive compulsive disorder, autistic disorder, and Asperger's disorder. The age range suitable for this assessment is 6 to 18 years of age for parent form (203-item) and the teacher form (204-item) and 8 to18 years of age for the self-report form (179-item). The 203-item parent form of CP-CBRS was used in this study and completed by the parents/primary caregivers of the participants. Total score for each subscale is expressed as T-score based on gender/age norms: T-scores range from 0-100. Higher score indicates higher severity. Lower score indicate lower severity.
Time Frame: Baseline, Week 60; Baseline, Week 252
Population: All enrolled participants who did not discontinue from the study for the reason 'Lost to follow up' at the first post-baseline observation and who had baseline and at least one post-baseline CP-CBRS assessment. No data was available for mixed episode due to not part of the statistical analysis plan..
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
T-score
  Manic Episode Week 60: number analyzed (Participants) | 102
  Manic Episode Week 60 | -7.09 (16.05)
  Manic Episode Week 252: number analyzed (Participants) | 20
  Manic Episode Week 252 | -14.85 (16.04)

25. Secondary Outcome: Mean Change From Baseline of Each Total Score CP-CBRS (DSM-IV-TR) ADHD Symptom Subscales (Hyperactive/Impulsive and Inattentive)
Description: as for outcome 24
Time Frame: Baseline, Week 12; Baseline, Week 60; Baseline, Week 252
Population: All enrolled participants who did not discontinue from the study for the reason 'Lost to follow up' at the first post-baseline observation and who had baseline and at least one post-baseline CP-CBRS assessment.
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
T Score
  Inattentive Week 12: number analyzed (Participants) | 205
  Inattentive Week 12 | -5.66 (13.44)
  Inattentive Week 60: number analyzed (Participants) | 102
  Inattentive Week 60 | -8.29 (14.59)
  Inattentive Week 252: number analyzed (Participants) | 20
  Inattentive Week 252 | -12.20 (13.32)
  Hyperactivity/Impulsivity Week 12: number analyzed (Participants) | 205
  Hyperactivity/Impulsivity Week 12 | -6.33 (13.44)
  Hyperactivity/Impulsivity Week 60: number analyzed (Participants) | 102
  Hyperactivity/Impulsivity Week 60 | -7.56 (14.65)
  Hyperactivity/Impulsivity Week 252: number analyzed (Participants) | 20
  Hyperactivity/Impulsivity Week 252 | -13.80 (15.66)

26. Secondary Outcome: Mean Change From Baseline of Each Total Score CP-CBRS DSM-IV-TR for Oppositional Defiant Disorder (ODD), Anxiety, Conduct Disorder and Major Depressive Episode
Description: as for outcome 24
Time Frame: Baseline, Week 12; Baseline, Week 60; Baseline, Week 252
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
T-score
  ODD Week 12: number analyzed (Participants) | 205
  ODD Week 12 | -1.77 (11.17)
  ODD Week 60: number analyzed (Participants) | 102
  ODD Week 60 | -1.65 (15.03)
  ODD Week 252: number analyzed (Participants) | 20
  ODD Week 252 | -5.15 (9.41)
  Anxiety Week 12: number analyzed (Participants) | 205
  Anxiety Week 12 | -3.36 (11.84)
  Anxiety Week 60: number analyzed (Participants) | 102
  Anxiety Week 60 | -4.00 (15.71)
  Anxiety Week 252: number analyzed (Participants) | 20
  Anxiety Week 252 | -12.00 (12.03)
  Conduct Disorder Week 12: number analyzed (Participants) | 205
  Conduct Disorder Week 12 | -2.12 (11.95)
  Conduct Disorder Week 60: number analyzed (Participants) | 102
  Conduct Disorder Week 60 | -1.97 (14.35)
  Conduct Disorder Week 252: number analyzed (Participants) | 20
  Conduct Disorder Week 252 | -2.65 (7.52)
  Major Depressive Episode Week 12: number analyzed (Participants) | 205
  Major Depressive Episode Week 12 | -3.31 (12.12)
  Major Depressive Episode Week 60: number analyzed (Participants) | 102
  Major Depressive Episode Week 60 | -3.43 (14.72)
  Major Depressive Episode Week 252: number analyzed (Participants) | 20
  Major Depressive Episode Week 252 | -9.05 (10.64)

27. Secondary Outcome: Mean Change From Baseline of Each Raw Score CP-CBRS Impairment Items Subscales for Schoolwork/Grades, Friendship/Relationships, and Home Life
Description: The Conners CBRS measures behaviors, emotions, and academic problems in children and adolescents. DSM-IV-TR symptom scales is included and assesses the following disorders: ADHD, conduct disorder, ODD, major depressive episode, manic episode, mixed episode, generalized anxiety disorder, separation anxiety disorder, social phobia, obsessive compulsive disorder, autistic disorder, and Asperger's disorder. The age range suitable for this assessment is 6 to 18 years of age for parent form (203-item) and the teacher form (204-item) and 8 to18 years of age for the self-report form (179-item). The 203-item parent form of CP-CBRS was used in this study and completed by the parents/primary caregivers of the participants. Schoolwork/grades, friendships/relationships, home life functioning scores range from 0=never to 3=very often. Raw scores are presented for each subscale with higher scores indicating higher severity and lower scores indicating lower severity.
Time Frame: Baseline, Week 12; Baseline, Week 60; Baseline, Week 252
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
units on a scale
  Schoolwork or Grades Week 12: number analyzed (Participants) | 205
  Schoolwork or Grades Week 12 | -0.35 (1.10)
  Schoolwork or Grades Week 60: number analyzed (Participants) | 102
  Schoolwork or Grades Week 60 | -0.48 (1.17)
  Schoolwork or Grades Week 252: number analyzed (Participants) | 20
  Schoolwork or Grades Week 252 | -0.65 (1.04)
  Friendships and relationships Week 12: number analyzed (Participants) | 205
  Friendships and relationships Week 12 | -0.23 (0.91)
  Friendships and relationships Week 60: number analyzed (Participants) | 102
  Friendships and relationships Week 60 | -0.26 (1.07)
  Friendships and relationships Week 252: number analyzed (Participants) | 20
  Friendships and relationships Week 252 | -0.70 (0.98)
  Home Life Week 12: number analyzed (Participants) | 205
  Home Life Week 12 | -0.30 (1.02)
  Home Life Week 60: number analyzed (Participants) | 102
  Home Life Week 60 | -0.48 (1.12)
  Home Life Week 252: number analyzed (Participants) | 20
  Home Life Week 252 | -0.80 (0.89)

28. Secondary Outcome: Mean Change From Baseline of Each Total Score CP-CBRS Content Subscale for Aggressive Behaviors, Academic Difficulties, Social Problems, and Violence Potential)
Description: CP-CBRS is a comprehensive assessment of a wide spectrum of behaviors, emotions, and academic problems in children and adolescents. It includes DSM-IV-TR symptom scales, empirical and rational scales, other clinical indicators and critical and impairment items. DSM-IV-TR symptom scales assess ADHD, conduct disorder, ODD, major depressive episode, manic episode, mixed episode, generalized anxiety disorder, separation anxiety disorder, social phobia, obsessive compulsive disorder, autistic disorder, and Asperger's disorder. The age range is 6 to 18 years of age for parent form (203-item) and the teacher form (204-item) and 8 to18 years of age self-report form (179-item). The parent form of Conners CBRS (CP-CBRS) was used in this study and completed by the parents/primary caregivers of the participants. Total score for each subscale is expressed as T-score based on gender/age norms: T-scores range from 0-100. Higher score indicates higher severity. Lower score indicate lower severity
Time Frame: Baseline, Week 12; Baseline, Week 60; Baseline, Week 252
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
T-score
  Aggressive behaviors Week 12: number analyzed (Participants) | 205
  Aggressive behaviors Week 12 | -1.53 (11.85)
  Aggressive behaviors Week 60: number analyzed (Participants) | 102
  Aggressive behaviors Week 60 | -0.80 (14.31)
  Aggressive behaviors Week 252: number analyzed (Participants) | 20
  Aggressive behaviors Week 252 | -5.65 (7.84)
  Academic difficulties Week 12: number analyzed (Participants) | 205
  Academic difficulties Week 12 | -4.39 (10.73)
  Academic difficulties Week 60: number analyzed (Participants) | 102
  Academic difficulties Week 60 | -4.37 (12.83)
  Academic difficulties Week 252: number analyzed (Participants) | 20
  Academic difficulties Week 252 | -8.55 (14.39)
  Social problems Week 12: number analyzed (Participants) | 205
  Social problems Week 12 | -0.37 (12.21)
  Social problems Week 60: number analyzed (Participants) | 102
  Social problems Week 60 | -1.12 (13.25)
  Social problems Week 252: number analyzed (Participants) | 20
  Social problems Week 252 | -4.65 (13.83)
  Violence Potential Week 12: number analyzed (Participants) | 205
  Violence Potential Week 12 | -1.25 (9.55)
  Violence Potential Week 60: number analyzed (Participants) | 102
  Violence Potential Week 60 | -0.79 (10.72)
  Violence Potential Week 252: number analyzed (Participants) | 20
  Violence Potential Week 252 | -3.70 (3.73)

29. Secondary Outcome: Mean Change From Baseline of the 5 Domain Scores Child Health and Illness Profile-Adolescent Edition (CHIP-AE) in 5 Health Outcome Domains (Satisfaction, Comfort, Resilience, Risk Avoidance and Achievement)
Description: CHIP-AE Child Report Form (CRF) is an adolescent rated assessment of their health status and level of functioning. The items in the 5 domains include: Achievement, Satisfaction, Comfort, Risk Avoidance, and Resilience. The majority of items assess frequency of activities or feelings using a 5-point response format (1=never, 5=always). Standard scores (T-scores) were established, with all domains and subdomains having a mean score of 50 and standard deviation of 10. Normative range is 40 to 60. Higher scores indicate better health and lower scores indicate worse health.
Time Frame: Baseline, Week 12; Baseline, Week 60; Baseline, Week 156
Population: All enrolled participants who did not discontinue from the study for the reason 'Lost to follow up' at the first post-baseline observation and who had baseline and at least one post-baseline CHIP-AE assessment.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
T-score
  Satisfaction Week 12: number analyzed (Participants) | 101
  Satisfaction Week 12 | 1.81 (6.86)
  Satisfaction Week 60: number analyzed (Participants) | 42
  Satisfaction Week 60 | 1.01 (7.62)
  Satisfaction Week 156: number analyzed (Participants) | 17
  Satisfaction Week 156 | 3.29 (5.52)
  Discomfort Week 12: number analyzed (Participants) | 100
  Discomfort Week 12 | 1.89 (4.88)
  Discomfort Week 60: number analyzed (Participants) | 41
  Discomfort Week 60 | 0.07 (5.65)
  Discomfort Week 156: number analyzed (Participants) | 16
  Discomfort Week 156 | 1.35 (7.29)
  Resilience Week 12: number analyzed (Participants) | 100
  Resilience Week 12 | -1.20 (8.85)
  Resilience Week 60: number analyzed (Participants) | 41
  Resilience Week 60 | -0.00 (8.69)
  Resilience Week 156: number analyzed (Participants) | 17
  Resilience Week 156 | 0.95 (8.26)
  Risk Avoidance Week 12: number analyzed (Participants) | 100
  Risk Avoidance Week 12 | 1.49 (6.26)
  Risk Avoidance Week 60: number analyzed (Participants) | 42
  Risk Avoidance Week 60 | -2.04 (6.17)
  Risk Avoidance Week 156: number analyzed (Participants) | 17
  Risk Avoidance Week 156 | -3.27 (5.81)
  Achievement Week 12: number analyzed (Participants) | 12
  Achievement Week 12 | 0.70 (5.86)
  Achievement Week 60: number analyzed (Participants) | 4
  Achievement Week 60 | -2.35 (8.40)
  Achievement Week 156: number analyzed (Participants) | 1
  Achievement Week 156 | 7.33 (NA) — Standard deviation was not calculated due to n=1.

30. Secondary Outcome: Mean Change From Baseline of the 5 Domain Scores Child Health and Illness Profile-Child Edition (CHIP-CE) in 5 Health Outcome Domains (Satisfaction, Comfort, Resilience, Risk Avoidance and Achievement)
Description: CHIP-CE Parent Report Form (PRF) is a parent rated assessment of a child's health status/level of functioning. The achievement domain describes developmentally appropriate role functioning in school and with peers. The majority of items assess frequency of activities or feelings using a 5-point response format (1=never, 5=always). Standard scores (T-scores) were established, with all domains and subdomains having a mean score of 50 and standard deviation of 10. Normative range is 40 to 60. Higher scores indicate better health and lower scores indicate worse health.
Time Frame: Baseline, Week 12; Baseline, Week 60; Baseline, Week 156
Population: All enrolled participants who did not discontinue from the study for the reason 'Lost to follow up' at the first post-baseline observation and who had baseline and at least one post-baseline CHIP-CE assessment.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
T-score
  Satisfaction Week 12: number analyzed (Participants) | 95
  Satisfaction Week 12 | 0.31 (8.65)
  Satisfaction Week 60: number analyzed (Participants) | 48
  Satisfaction Week 60 | -1.87 (9.49)
  Satisfaction Week 156: number analyzed (Participants) | 12
  Satisfaction Week 156 | -1.74 (5.34)
  Discomfort Week 12: number analyzed (Participants) | 96
  Discomfort Week 12 | -0.22 (8.43)
  Discomfort Week 60: number analyzed (Participants) | 48
  Discomfort Week 60 | -2.89 (12.11)
  Discomfort Week 156: number analyzed (Participants) | 12
  Discomfort Week 156 | -0.09 (9.37)
  Resilience Week 12: number analyzed (Participants) | 95
  Resilience Week 12 | 0.58 (10.93)
  Resilience Week 60: number analyzed (Participants) | 48
  Resilience Week 60 | -1.07 (12.09)
  Resilience Week 156: number analyzed (Participants) | 12
  Resilience Week 156 | 0.83 (9.33)
  Risk Avoidance and Achievement Week 12: number analyzed (Participants) | 96
  Risk Avoidance and Achievement Week 12 | 1.54 (8.10)
  Risk Avoidance and Achievement Week 60: number analyzed (Participants) | 48
  Risk Avoidance and Achievement Week 60 | 1.89 (8.95)
  Risk Avoidance and Achievement Week 156: number analyzed (Participants) | 12
  Risk Avoidance and Achievement Week 156 | 4.49 (13.89)
  Achievement Week 12: number analyzed (Participants) | 96
  Achievement Week 12 | 2.75 (9.01)
  Achievement Week 60: number analyzed (Participants) | 48
  Achievement Week 60 | 2.92 (10.58)
  Achievement Week 156: number analyzed (Participants) | 12
  Achievement Week 156 | 4.28 (9.54)

31. Secondary Outcome: Mean Change From Baseline of Total Score Euro-Qol Questionnaire - 5 Dimensions 3 Levels (EQ-5D-3L) Health State for Parent
Description: The EQ-5D-3L is a generic, multidimensional, health-related, quality-of-life (QoL) instrument that contains 2 parts: a health status profile and a visual analog scale to rate global health-related QoL. The profile allows respondents to rate their health state in 5 health dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels of measure: no problems, some problems, and severe problems. The 5 dimensions of the health state profile are reported as a population-based (UK or US) health index score of theoretically possible health states ranging from 0-1; where 0 is death and 1 is perfect health. i.e., higher is better. Parents of the participants completed the EQ-5D-3L form for rating their own quality of life.
Time Frame: Baseline, Week 12; Baseline, Week 60; Baseline, Week 252
Population: Parents of the participants completed the EQ-5D-3L form for rating their own quality of life, for parents of participants who did not discontinue from the study for the reason 'Lost to follow up' at the first post-baseline observation and who had baseline and at least one post-baseline EQ-5D-3L VAS assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
units on a scale
  UK population-based Week 12: number analyzed (Participants) | 129
  UK population-based Week 12 | -0.011 (0.194)
  UK population-based Week 60: number analyzed (Participants) | 64
  UK population-based Week 60 | -0.016 (0.203)
  UK population-based Week 252: number analyzed (Participants) | 15
  UK population-based Week 252 | 0.008 (0.087)
  US population-based Week 12: number analyzed (Participants) | 129
  US population-based Week 12 | -0.009 (0.140)
  US population-based Week 60: number analyzed (Participants) | 64
  US population-based Week 60 | -0.014 (0.144)
  US population-based Week 252: number analyzed (Participants) | 15
  US population-based Week 252 | 0.019 (0.077)

32. Secondary Outcome: Mean Change From Baseline of Total Score EQ-5D-3L Visual Analog Scale (VAS) for Parent
Description: The EQ-5D-3L is a generic, multidimensional, health-related, QoL instrument that contains 2 parts: a health status profile and a visual analog scale to rate global health-related QoL. The visual analog scale reported records the respondent's self-rated health state on a vertical line where the endpoints are labeled 100 being "best imaginable health state" and 0 being "worst imaginable health state." Parents of the participants complete EQ-5D-3L form for rating their own health.
Time Frame: Baseline, Week 12; Baseline, Week 60; Baseline, Week 252
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
units on a scale
  Week 12: number analyzed (Participants) | 129
  Week 12 | -0.845 (21.908)
  Week 60: number analyzed (Participants) | 63
  Week 60 | 2.968 (20.800)
  Week 252: number analyzed (Participants) | 15
  Week 252 | 2.467 (14.252)

33. Secondary Outcome: Mean Change of From Baseline Total Score EQ-5D-3L Health State for Child
Description: The EQ-5D-3L is a generic, multidimensional, health-related, QoL instrument that contains 2 parts: a health status profile and a visual analog scale to rate global health-related QoL. The profile allows respondents to rate their health state in 5 health dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels of measure: no problems, some problems, and severe problems. The 5 dimensions of the health state profile are reported as a population-based (UK or US) health index score of theoretically possible health states ranging from 0-1; where 0 is death and 1 is perfect health. Parents of the participants aged 6 to 11 years completed the EQ-5D-3L form regarding the participants health-related quality of life. i.e., young children were unable to assess their own quality of life so the parents assessed the child's quality of life for them.
Time Frame: Baseline, Week 12; Baseline, Week 60; Baseline, Week 252
Population: All enrolled participants who did not discontinue from the study for the reason 'Lost to follow up' at the first post-baseline observation and who had baseline and at least one post-baseline EQ-5D-3L assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
units on a scale
  UK population based Week 12: number analyzed (Participants) | 72
  UK population based Week 12 | 0.024 (0.132)
  UK population based Week 60: number analyzed (Participants) | 38
  UK population based Week 60 | 0.010 (0.138)
  UK population based Week 252: number analyzed (Participants) | 3
  UK population based Week 252 | 0.000 (0.000)
  US population based Week 12: number analyzed (Participants) | 72
  US population based Week 12 | 0.019 (0.109)
  US population based Week 60: number analyzed (Participants) | 38
  US population based Week 60 | 0.006 (0.109)
  US population based Week 252: number analyzed (Participants) | 3
  US population based Week 252 | 0.000 (0.000)

34. Secondary Outcome: Mean Change of From Baseline Total Score EQ-5D-3L VAS for Child
Description: EQ-5D-3L is a generic, multidimensional, health-related, QoL instrument that contains 2 parts: a health status profile and a visual analog scale to rate global health-related QoL. The visual analog scale reported records the respondent's self-rated health state on a vertical line where the endpoints are labeled 100 being "best imaginable health state" and 0 being "worst imaginable health state." Parents of the participants aged 6 to 11 years complete the EQ-5D-3L form for rating the participants health-related QoL, EQ-5D-3L. i.e., the young child was unable to assess their own quality of life then the parent assessed the child's quality of life.
Time Frame: Baseline, Week 12; Baseline, Week 60; Baseline, Week 252
Population: All enrolled participants who did not discontinue from the study for the reason 'Lost to follow up' at the first post-baseline observation and who had baseline and at least one post-baseline EQ-5D-3L VAS assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
units on a scale
  Week 12: number analyzed (Participants) | 72
  Week 12 | -2.389 (21.636)
  Week 60: number analyzed (Participants) | 38
  Week 60 | 2.842 (15.023)
  Week 252: number analyzed (Participants) | 3
  Week 252 | -1.667 (2.887)

35. Secondary Outcome: Mean Change From Baseline of Total Score EQ-5D-3L Health State for Adolescent
Description: EQ-5D-3L is a generic, multidimensional, health-related, QoL instrument that contains 2 parts: a health status profile and a visual analog scale to rate global health-related QoL. The profile allows respondents to rate their health state in 5 health dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels of measure: no problems, some problems, and severe problems. The 5 dimensions of the health state profile are reported as a population-based (UK or US) health index score of theoretically possible health states ranging from 0-1; where 0 is death and 1 is perfect health. i.e., higher is better. Participants aged 12 years or older rate their own health-related quality of life using EQ-5D-3L.
Time Frame: Baseline, Week 12; Baseline, Week 60; Baseline, Week 252
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
units on a scale
  UK population based Week 12: number analyzed (Participants) | 106
  UK population based Week 12 | -0.010 (0.122)
  UK population based Week 60: number analyzed (Participants) | 50
  UK population based Week 60 | -0.016 (0.217)
  UK population based Week 252: number analyzed (Participants) | 10
  UK population based Week 252 | 0.008 (0.055)
  US population based Week 12: number analyzed (Participants) | 106
  US population based Week 12 | -0.008 (0.101)
  US population based Week 60: number analyzed (Participants) | 50
  US population based Week 60 | -0.005 (0.150)
  US population based Week 252: number analyzed (Participants) | 10
  US population based Week 252 | 0.013 (0.053)

36. Secondary Outcome: Mean Change From Baseline of Total Score EQ-5D-3L VAS
Description: EQ-5D-3L is a generic, multidimensional, health-related, QoL instrument that contains 2 parts: a health status profile and a visual analog scale to rate global health-related QoL. The visual analog scale reported records the respondent's self-rated health state on a vertical line where the endpoints are labeled 100 being "best imaginable health state" and 0 or being "worst imaginable health state." Participants aged 12 years or older rated their own health-related quality of life using the EQ-5D-3L VAS scale.
Time Frame: Baseline, Week 12; Baseline, Week 60; Baseline, Week 252
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edivoxetine
Number analyzed (Participants) | 264
units on a scale
  Week 12: number analyzed (Participants) | 107
  Week 12 | 2.364 (21.224)
  Week 60: number analyzed (Participants) | 50
  Week 60 | 1.620 (18.025)
  Week 252: number analyzed (Participants) | 10
  Week 252 | 1.200 (12.007)

37. Secondary Outcome: Mean Change From Baseline of Total Score Woodcock Johnson III Test of Achievement ([WJ III ACH])
Description: The Woodcock Johnson (WJ III ACH) (Woodcock 2001) is designed to measure academic achievement and evaluates a person aged 2 to 90 years and the tool takes 60 to 160 minutes to complete depending on a person's academic level. The WJ III ACH has 2 parallel forms (A and B) that can be administered in an alternating fashion. The WCJ III ACH uses standard scores (Deviation IQ) with an average standard score of 100 and a standard deviation of 15. Higher scores indicate better abilities/achievements. Lower scores indicate worse abilities/achievements.
Time Frame: Baseline, Week 60
Population: All enrolled participants with baseline and at least one post-baseline WJ III ACH assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edivoxetine
Number analyzed (Participants) | 20
units on a scale | 0.05 (5.01)

38. Secondary Outcome: Mean Change From Baseline of Total Score Wide Range Achievement Test (WRAT 4)
Description: The WRAT 4 is a norm-referenced test that measures the basic academic skills of word reading, sentence comprehension, spelling, and math computation. There are 2 alternate forms (Blue Form, Green Form) that can be used interchangeably with comparable results. It can be used to evaluate a person aged 5 to 94 years and the administration time is 30 to 45 minutes for children (8 years or older) and adults, and 15 to 25 minutes for young children (ages 5 to 7 years). The age-normed standard scores range from 55 - 145 and for each subtest/composite includes word reading, sentence comprehension, spelling, math computation and reading composite. Higher scores indicate better abilities/achievements. Lower scores indicate worse abilities/achievements.
Time Frame: Baseline, Week 60
Population: All enrolled participants with baseline and at least one post-baseline WRAT 4 assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edivoxetine
Number analyzed (Participants) | 10
units on a scale
  Word Reading | -3.30 (25.84)
  Sentence Comprehension | -1.80 (25.94)
  Spelling | -6.40 (22.08)
  Math Computation | -8.50 (25.21)
  Reading Composite | 16.20 (36.10)

39. Secondary Outcome: Mean Change From Baseline of Total Score Wechsler Intelligence Scale for Children Fourth Edition (WISC-IV)
Description: The fourth edition of the WISC assessment (WISC-IV®) is administered to children ranging from 6 years to 16 years, 11 months. It contains 10 core subtests and 5 supplementary subtests, and takes 65-80 minutes to complete. In this study, Digit Span and Letter-Number Sequencing subtests were completed. Scaled scores range from 1 to 19. Higher scores denote better performance. Lower scores denote worse performance.
Time Frame: Baseline, Week 60
Population: All enrolled participants with baseline and at least one post-baseline WISC-IV assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edivoxetine
Number analyzed (Participants) | 72
units on a scale
  Digit Span Scaled Score | 0.61 (2.42)
  Letter-Number Sequencing Scaled Score | 0.63 (2.53)

40. Secondary Outcome: Mean Change From Baseline of Total Score Wechsler Adult Intelligence Scale - Third Edition (WAIS-III)
Description: The WAIS-III® was used in the participants aged 17 years or older. Comprehensive reporting on the participant's intellectual ability is not required in this study. Raw scores for each of the 14 subtests are reported. Raw score ranges for each subtest are as follows: picture completion (0-25), vocabulary (0-66), digit symbol coding (0-133), similarities (0-33), block design (0-68), arithmetic (0-22), matrix reasoning (0-26), digit span forward and backward total (0-30), information (0-28), picture arrangement (0-22), comprehension (0-33), symbol search (0-60), letter-number sequencing (0-21), and object assembly (0-52). Higher scores reflect better performance and lower scores reflect lower performance.
Time Frame: Baseline, Week 60
Population: All enrolled participants with baseline and at least one post-baseline WAIS-III assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edivoxetine
Number analyzed (Participants) | 2
units on a scale
  Picture Completion | 0.50 (0.71)
  Vocabulary | -11.50 (12.02)
  Digit-Symbol Coding | -22.00 (39.60)
  Similarities | 4.00 (7.07)
  Block Design | -8.00 (29.70)
  Arithmetic | 6.00 (9.90)
  Matrix Reasoning | 3.50 (2.12)
  Digit Span | 4.00 (2.83)
  Information | 3.50 (2.12)
  Picture Arrangement | -2.50 (0.71)
  Comprehension | -9.00 (11.31)
  Symbol Search | -5.00 (7.07)
  Letter Number Sequencing | 7.50 (12.02)
  Object Assembly | -10.00 (18.38)

ADVERSE EVENTS:
Time Frame: Overall edivoxetine treatment adverse event data were collected for up to 5 years.
Description: 264 participants are the evaluable participants defined as enrolled participants who did not discontinue from the study for the reason 'Lost to follow up' at the first post-baseline observation.
Groups:
- Edivoxetine (Open-Label): Edivoxetine: 0.1 mg/kg/day or participant specific known stable dose (rollover participants) up to 0.3 mg/kg/day, oral, daily for up to 5 years.
- Edivoxetine (Follow Up): The follow up period is an optional taper of Edivoxetine. Treatment may be tapered or discontinued, over a period of 10 to 18 days.
Arm/Group | Edivoxetine (Open-Label) | Edivoxetine (Follow Up)
Serious Adverse Events (participants affected / at risk) | 7/264 | 1/80
Other Adverse Events (participants affected / at risk) | 155/264 | 5/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edivoxetine (Open-Label) (N=264) | Edivoxetine (Follow Up) (N=80)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intentional product misuse (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edivoxetine (Open-Label) (N=264) | Edivoxetine (Follow Up) (N=80)
Abdominal pain upper (Gastrointestinal disorders) | 22 (28) | 2 (2)
Nausea (Gastrointestinal disorders) | 35 (48) | 0 (0)
Vomiting (Gastrointestinal disorders) | 45 (69) | 0 (0)
Fatigue (General disorders) | 16 (19) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 15 (17) | 0 (0)
Nasopharyngitis (Infections and infestations) | 18 (28) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 15 (19) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 35 (44) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 15 (16) | 1 (1)
Headache (Nervous system disorders) | 45 (61) | 0 (0)
Somnolence (Nervous system disorders) | 14 (15) | 0 (0)
Irritability (Psychiatric disorders) | 22 (22) | 0 (0)

LIMITATIONS AND CAVEATS:
Terminated due to low 5 year completer number and not meeting primary objective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days